CLINICAL TRIAL: NCT05729672
Title: Developing and Testing a Small Private Online Course (SPOC) for Nurse-patient Communication About Sex.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jian Tao Lee, Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 106-2629-S-182-002
Record Dates: First submitted 2022-12-29; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Nurse-Patient Relations
Keywords: sex education; gender-sensitivity; nurse-patient communication; continuing education; SPOC

STUDY DESIGN:
Intervention Model Description: The course includes five online teaching and learning modules and two hours of offline teaching and learning, using MOOCs/SPOCs online teaching system and constructs on the Chinese Open Education platform. For this prospective, randomized controlled trial, 150 nurses working in a medical center in northern Taiwan were recruited and randomized into 2 groups. The experimental group (n=75) received the Nightingale in Gen-sEx course. The control group (n=75) received without course. Data were collected at baseline, 1month, and 3 months after the course.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (Experimental): The experimental group will participate in the SPOC- based education program, consisting of five online teaching and learning modules over the span of 3 months and two hours of offline classroom.
  Interventions: Behavioral: Received the Nightingale in Gen-sEx course
- The control group (No Intervention): The control group will not receive any education. Data will be collected at baseline, 1 month and 3 months after intervention.

INTERVENTIONS:
Behavioral: Received the Nightingale in Gen-sEx course — The experimental group (n=75) will participate in the SPOC- based education program, consisting of five online teaching and learning modules over the span of 3 months and two hours of offline classroom.
  Arms: The experimental group

SUMMARY:
This is a three-year research project. The goal is to develop and test "The SPOC-based blended teaching and learning platform (Nightingale in Gen-sEx)" that integrates effective educational strategies and e-learning methods to meet the Taiwanese nurse's learning needs. This project is aimed at resolving sexual education learning problems in nursing continuing education due to the time constraints at clinical sites and the shortage of teaching staff. Nurse-patient communication attitudes and skills about sex will be enhanced.

DETAILED DESCRIPTION:
The research team constructed a course for hospital nurses that followed the commonly used ADDIE (Analysis, Design, Development, Implementation, and Evaluation) model. The first year research purpose is to: (1) explore the characteristics of nursing-patient communication about sex and the core educational needs content for nurses using triangulation methods. (2) Construct gender-sensitivity structures characteristics of nursing-patient communication about sex and course framework according to the modified Delphi method results and course needs assessment. The second year develops the SPOC-based blended teaching and learning platform (E-generation Angel of Happiness") and conducts a pilot study to test and correct the course content and method. In the third year a pretest-posttest randomized control group design will be implemented to investigate the effectiveness of the course "E-generation Angel of Happiness" in improving competencies of nurse-patient communication about sex, including attitudes, and practices, among nurses.

ELIGIBILITY:
Inclusion Criteria:

1. 20 to 50 years old.
2. Below N3 rank.
3. Full-time nurse in clinical care.
4. Have smartphones or computers, and be able to use and be online.
5. Nurses who are willing to participate in this study and sign the consent form

Exclusion Criteria:

1. Will leave within 3 months.
2. unable to learn online.
3. The working units are surgery room, recovery room, hospice ward, supply center.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2020-08-16 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Sexual Communication between Nurses and Patients | Data were collected at baseline.
  The research project assessed changes in sexual communication between Nurses and Patients by Sexual Communication Scale between Nurses and Patients(SCS-NS) from baseline to 3 months after the course.
  Sexual Communication Scale between Nurses and Patients (SCS-NS) is developed with reference to "Questionnaires of barriers to discussing sexuality with patients" by Hordern et al. (2009). It has 14 items and consists of two parts: 1. Frequency of sexual communication with patients (4 items ) and 2. Sexual Communication Barrier Scale (10 questions). The Sexual Communication Obstacle Scale adopts a Likert 5-point scale for scoring, and the higher the score, the higher the sexual barrier to talking with the patient and the lower the level of nurse-patient communication. The questionnaire will undergo expert validity testing again, and the internal consistency of the scale reliability will be evaluated by the Cronbach Alpha coefficient.
Sexual Communication between Nurses and Patients | Data were collected at 1 month after the course.
  The research project assessed changes in sexual communication between Nurses and Patients by Sexual Communication Scale between Nurses and Patients(SCS-NS) from baseline to 3 months after the course.
  Sexual Communication Scale between Nurses and Patients (SCS-NS) is developed with reference to "Questionnaires of barriers to discussing sexuality with patients" by Hordern et al. (2009). It has 14 items and consists of two parts: 1. Frequency of sexual communication with patients (4 items ) and 2. Sexual Communication Barrier Scale (10 questions). The Sexual Communication Obstacle Scale adopts a Likert 5-point scale for scoring, and the higher the score, the higher the sexual barrier to talking with the patient and the lower the level of nurse-patient communication. The questionnaire will undergo expert validity testing again, and the internal consistency of the scale reliability will be evaluated by the Cronbach Alpha coefficient.
Sexual Communication between Nurses and Patients | Data were collected at 3 month after the course.
  The research project assessed changes in sexual communication between Nurses and Patients by Sexual Communication Scale between Nurses and Patients(SCS-NS) from baseline to 3 months after the course.
  Sexual Communication Scale between Nurses and Patients (SCS-NS) is developed with reference to "Questionnaires of barriers to discussing sexuality with patients" by Hordern et al. (2009). It has 14 items and consists of two parts: 1. Frequency of sexual communication with patients (4 items ) and 2. Sexual Communication Barrier Scale (10 questions). The Sexual Communication Obstacle Scale adopts a Likert 5-point scale for scoring, and the higher the score, the higher the sexual barrier to talking with the patient and the lower the level of nurse-patient communication. The questionnaire will undergo expert validity testing again, and the internal consistency of the scale reliability will be evaluated by the Cronbach Alpha coefficient.
Gender sensitivity | Data were collected at baseline.
  The research project assessed changes in gender sensitivity by Gender-Sensitivity Scale for Nurses from baseline to 3 months after the course.
  The scale" Gender-Sensitivity Scale for Nurses" is a self-development scale, referring to the gender-blind connotation of sexual health guidance for medical staff proposed by Lee et al. (2017) and the Gender Awareness Scale developed by Verdonk et al. (Njmegen Medical Gender Awareness Scale). (2007), to be developed. The scale consists of 14 items, with a five-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Questions 10, 12, 13, and 14 are reverse-scoring, and the scoring range is 10-50 points. The higher the score, the lower the gender sensitivity and gender blindness. The questionnaire will undergo the expert validity test, and Cronbach's α coefficient will evaluate the internal consistency of the scale reliability. In this study, Cronbach's alpha for the quantitative learning needs assessment was 0.79.
Gender sensitivity | Data were collected at 1 month after the course.
  The research project assessed changes in gender sensitivity by Gender-Sensitivity Scale for Nurses from baseline to 3 months after the course.
  The scale" Gender-Sensitivity Scale for Nurses" is a self-development scale, referring to the gender-blind connotation of sexual health guidance for medical staff proposed by Lee et al. (2017) and the Gender Awareness Scale developed by Verdonk et al. (Njmegen Medical Gender Awareness Scale). (2007), to be developed. The scale consists of 14 items, with a five-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Questions 10, 12, 13, and 14 are reverse-scoring, and the scoring range is 10-50 points. The higher the score, the lower the gender sensitivity and gender blindness. The questionnaire will undergo the expert validity test, and Cronbach's α coefficient will evaluate the internal consistency of the scale reliability. In this study, Cronbach's alpha for the quantitative learning needs assessment was 0.79.
Gender sensitivity | Data were collected at 3 month after the course.
  The research project assessed changes in gender sensitivity by Gender-Sensitivity Scale for Nurses from baseline to 3 months after the course.
  The scale" Gender-Sensitivity Scale for Nurses" is a self-development scale, referring to the gender-blind connotation of sexual health guidance for medical staff proposed by Lee et al. (2017) and the Gender Awareness Scale developed by Verdonk et al. (Njmegen Medical Gender Awareness Scale). (2007), to be developed. The scale consists of 14 items, with a five-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Questions 10, 12, 13, and 14 are reverse-scoring, and the scoring range is 10-50 points. The higher the score, the lower the gender sensitivity and gender blindness. The questionnaire will undergo the expert validity test, and Cronbach's α coefficient will evaluate the internal consistency of the scale reliability. In this study, Cronbach's alpha for the quantitative learning needs assessment was 0.79.

SECONDARY OUTCOMES:
Sexual health care attitudes | Data were collected at baseline, 1 month, and 3 months after the course.
  The research project assessed changes in sexual health care attitude by the Sexual Health Care Scale-Attitude (SHCS-A) from baseline to 3 months after the course.
  The Sexual Health Care Scale-Attitude (SHCS-A) was used to measure attitudes toward Sexual Health Care for oncology patients. This scale was developed for oncology nurses, and has been proven valid and reliable (Kim & Kim, 2011). The scale consists of 17 items, with each item rated on a three-point scale ranging from 1 (agree) to 3 (disagree). The total scores range from 17 to 51. The SHCS-A consists of four factors: discomfort in providing SHC, feeling uncertain about patient's acceptance, fear of colleagues' negative response, and lack of environmental support. Higher scores indicate a more positive attitude toward SHC for oncology patients. Cronbach's α for this scale was .93 (Kim & Kim, 2011).
Readiness of talking about sex | Data were collected at baseline, 1 month, and 3 months after the course.
  The research project assessed changes in readiness of talking about sex by Lee's (2019) "Readiness to Talk About Sex Stage Scale" from baseline to 3 months after the course.
  Lee's (2019) "Readiness to Talk About Sex Stage Scale" assesses nurses' readiness to talk about sex with patients: "I do not think it is necessary to talk to patients about sex or provide sexual health information"; "I do not want to talk about sex with patients, nor have I talking to patients about sex"; "I think I should give sexual health advice to patients or talk to patients about sex, but I do not want to do so yet"; "I want to talk to patients about sex or provide sexual health counseling, however, I still not started"; "I have started talking to patients about sex or giving sexual health counseling"; "I have started talking to patients' about sex or giving sexual health counseling and have done so routinely for more than three months'"; and according to These five options are scored on a scale of 1 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Tao LEE, Professor, Principal Investigator — Chang Gung University
Locations (1):
- Cheng Gung Memorial Hospital, Taoyuan District, Guishan Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aloush SM. Lecture-based education versus simulation in educating student nurses about central line-associated bloodstream infection-prevention guidelines. J Vasc Nurs. 2019 Jun;37(2):125-131. doi: 10.1016/j.jvn.2018.11.006. Epub 2019 Jan 7. PMID 31155159
- [Background] Annerstedt CF, Glasdam S. Nurses' attitudes towards support for and communication about sexual health-A qualitative study from the perspectives of oncological nurses. J Clin Nurs. 2019 Oct;28(19-20):3556-3566. doi: 10.1111/jocn.14949. Epub 2019 Jun 4. PMID 31165516
- [Background] Bardach, L., Rushby, J. V., Kim, L. E., & Klassen, R. M. (2021). Using video-and text-based situational judgement tests for teacher selection: a quasi-experiment exploring the relations between test format, subgroup differences, and applicant reactions. European Journal of Work and Organizational Psychology, 30(2), 251-264. doi: 10.1080/1359432X.2020.1736619
- [Background] Button D, Harrington A, Belan I. E-learning & information communication technology (ICT) in nursing education: A review of the literature. Nurse Educ Today. 2014 Oct;34(10):1311-23. doi: 10.1016/j.nedt.2013.05.002. Epub 2013 Jun 18. PMID 23786869
- [Background] Cant RP, Cooper SJ. Simulation-based learning in nurse education: systematic review. J Adv Nurs. 2010 Jan;66(1):3-15. doi: 10.1111/j.1365-2648.2009.05240.x. PMID 20423432
- [Background] Delen, E., Liew, J., & Willson, V. (2014). Effects of interactivity and instructional scaffolding on learning: Self-regulation in online video-based environments. Computers & Education, 78, 312-320.
- [Background] Faulder GS, Riley SC, Stone N, Glasier A. Teaching sex education improves medical students' confidence in dealing with sexual health issues. Contraception. 2004 Aug;70(2):135-9. doi: 10.1016/j.contraception.2004.03.010. PMID 15288218
- [Background] Fennell R, Grant B. Discussing sexuality in health care: A systematic review. J Clin Nurs. 2019 Sep;28(17-18):3065-3076. doi: 10.1111/jocn.14900. Epub 2019 Jun 13. PMID 31017326
- [Background] Frederick NN, Campbell K, Kenney LB, Moss K, Speckhart A, Bober SL. Barriers and facilitators to sexual and reproductive health communication between pediatric oncology clinicians and adolescent and young adult patients: The clinician perspective. Pediatr Blood Cancer. 2018 Aug;65(8):e27087. doi: 10.1002/pbc.27087. Epub 2018 Apr 26. PMID 29697189
- [Background] Habes EV, Jepma P, Parlevliet JL, Bakker A, Buurman BM. Video-based tools to enhance nurses' geriatric knowledge: A development and pilot study. Nurse Educ Today. 2020 Jul;90:104425. doi: 10.1016/j.nedt.2020.104425. Epub 2020 Apr 3. PMID 32311666
- [Background] Huang CY, Tsai LY, Liao WC, Lee S. Nursing interventions on sexual health: validation of the NISH Scale in baccalaureate nursing students in Taiwan. J Sex Med. 2012 Oct;9(10):2600-8. doi: 10.1111/j.1743-6109.2012.02784.x. Epub 2012 May 22. PMID 22616685
- [Background] Jonsdottir JI, Zoega S, Saevarsdottir T, Sverrisdottir A, Thorsdottir T, Einarsson GV, Gunnarsdottir S, Fridriksdottir N. Changes in attitudes, practices and barriers among oncology health care professionals regarding sexual health care: Outcomes from a 2-year educational intervention at a University Hospital. Eur J Oncol Nurs. 2016 Apr;21:24-30. doi: 10.1016/j.ejon.2015.12.004. Epub 2016 Jan 5. PMID 26952675
- [Background] Kim JH, Shin JS. Effects of an online problem-based learning program on sexual health care competencies among oncology nurses: a pilot study. J Contin Educ Nurs. 2014 Sep;45(9):393-401. doi: 10.3928/00220124-20140826-02. PMID 25153429
- [Background] McDonald EW, Boulton JL, Davis JL. E-learning and nursing assessment skills and knowledge - An integrative review. Nurse Educ Today. 2018 Jul;66:166-174. doi: 10.1016/j.nedt.2018.03.011. Epub 2018 Mar 21. PMID 29705504
- [Background] Mohamadi-Bolbanabad S, Farnam F, Pakgohar M. The Effect of Virtual Education on Midwifery Students' Knowledge of Child Sexual Training. Iran J Nurs Midwifery Res. 2019 Sep-Oct;24(5):337-342. doi: 10.4103/ijnmr.IJNMR_96_18. PMID 31516518
- [Background] Percat A, Elmerstig E. "We should be experts, but we're not": Sexual counselling at the antenatal care clinic. Sex Reprod Healthc. 2017 Dec;14:85-90. doi: 10.1016/j.srhc.2017.10.001. Epub 2017 Oct 12. PMID 29195640
- [Background] Quinn C, Platania-Phung C, Bale C, Happell B, Hughes E. Understanding the current sexual health service provision for mental health consumers by nurses in mental health settings: Findings from a Survey in Australia and England. Int J Ment Health Nurs. 2018 Oct;27(5):1522-1534. doi: 10.1111/inm.12452. Epub 2018 Mar 25. PMID 29575550
- [Background] Quinn GP, Bowman Curci M, Reich RR, Gwede CK, Meade CD; ENRICH/ECHO Working Group; Vadaparampil ST. Impact of a web-based reproductive health training program: ENRICH (Educating Nurses about Reproductive Issues in Cancer Healthcare). Psychooncology. 2019 May;28(5):1096-1101. doi: 10.1002/pon.5063. Epub 2019 Apr 5. PMID 30882960
- [Background] Reese JB, Lepore SJ, Daly MB, Handorf E, Sorice KA, Porter LS, Tulsky JA, Beach MC. A brief intervention to enhance breast cancer clinicians' communication about sexual health: Feasibility, acceptability, and preliminary outcomes. Psychooncology. 2019 Apr;28(4):872-879. doi: 10.1002/pon.5036. Epub 2019 Mar 13. PMID 30811732
- [Background] Ross MW, Leshabari S, Rosser BRS, Trent M, Mgopa L, Wadley J, Kohli N, Agardh A. Evaluation of an assessment instrument for a sexual health curriculum for nurses and midwifery students in Tanzania: The sexual health education for professionals scale (SHEPS). Appl Nurs Res. 2018 Apr;40:152-156. doi: 10.1016/j.apnr.2018.01.005. Epub 2018 Feb 1. PMID 29579491
- [Background] Sung SC, Lin YC. Effectiveness of the sexual healthcare education in nursing students' knowledge, attitude, and self-efficacy on sexual healthcare. Nurse Educ Today. 2013 May;33(5):498-503. doi: 10.1016/j.nedt.2012.06.019. Epub 2012 Jul 10. PMID 22789872
- [Background] Tsai YF. Nurses' facilitators and barriers for taking a sexual history in Taiwan. Appl Nurs Res. 2004 Nov;17(4):257-64. doi: 10.1016/j.apnr.2004.09.011. PMID 15573334
- [Background] Vural, O. F. (2013). The Impact of a Question-Embedded Video-Based Learning Tool on E-Learning. Educational Sciences: Theory and Practice, 13(2), 1315-1323.
- [Background] Wang LY, Pierdomenico A, Lefkowitz A, Brandt R. Female Sexual Health Training for Oncology Providers: New Applications. Sex Med. 2015 Sep;3(3):189-97. doi: 10.1002/sm2.66. Epub 2015 Apr 14. PMID 26468382
- [Background] Webb L, Clough J, O'Reilly D, Wilmott D, Witham G. The utility and impact of information communication technology (ICT) for pre-registration nurse education: A narrative synthesis systematic review. Nurse Educ Today. 2017 Jan;48:160-171. doi: 10.1016/j.nedt.2016.10.007. Epub 2016 Oct 26. PMID 27816862
- [Background] World Health Organization (2017). Sexual and Reproductive Health, Retrieved from http://www.who.int.proxy.lib.cgu.edu.tw:81/reproductivehealth/topics/sexual_health/sh_definitions/en/
- [Background] Zhang, D., Zhou, L., Briggs, R. O., & Nunamaker Jr, J. F. (2006). Instructional video in e-learning: Assessing the impact of interactive video on learning effectiveness. Information & management, 43(1), 15-27. doi: 10.1016/j.im.2005.01.004